CLINICAL TRIAL: NCT04813120
Title: The Use of a New Digital Mirror Therapy System Providing Unilateral and Bilateral Mirror Visual Feedback for Patients With Stroke: Treatment Effects and EEG-physiological Evidence
Brief Title: Digital Mirror Therapy With Uni- and Bilateral Mirror Visual Feedback After Stroke: Treatment Effects and EEG Evidence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 202002234A3
Record Dates: First submitted 2021-03-21; First posted 2021-03-24 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2023-08

CONDITIONS: Stroke; Cerebrovascular Disorders; Central Nervous System Diseases
Keywords: digital rehabilitation; cerebrovascular accident; mirror visual feedback; brain electrophysiology
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Central Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Uni-MVF condition and unimanual training mode using the new MT system (UM-UT) (Experimental): The following common categories of upper-limb movements and actions will be selected and included in this group: (a) active range of motion (AROM) exercises, (b) reaching movements, and (c) object manipulation.
  Interventions: Behavioral: Uni-MVF condition and unimanual training mode using the new MT system (UM-UT)
- Uni-MVF condition and bimanual training mode using the new MT system (UM-BT) (Experimental): The following common categories of upper-limb movements and actions will be selected and included in this group: (a) active range of motion (AROM) exercises, (b) reaching movements, and (c) object manipulation.
  Interventions: Behavioral: Uni-MVF condition and bimanual training mode using the new MT system (UM-BT)
- Bi-MVF condition and bimanual training mode using the new MT system (BM-BT) (Experimental): The following common categories of upper-limb movements and actions will be selected and included in this group: (a) active range of motion (AROM) exercises, (b) reaching movements, and (c) object manipulation.
  Interventions: Behavioral: Bi-MVF condition and bimanual training mode using the new MT system (BM-BT)
- Traditional MT using a mirror box (Active Comparator): The following common categories of upper-limb movements and actions will be selected and included in this group: (a) active range of motion (AROM) exercises, (b) reaching movements, and (c) object manipulation.
  Interventions: Behavioral: Traditional MT using a mirror box

INTERVENTIONS:
Behavioral: Uni-MVF condition and unimanual training mode using the new MT system (UM-UT) — For the UM-UT group, the participants will be seated in front of the new MT system, and will be instructed to watch the real-time image reflection of movements of the non-affected arm and hand on the screen carefully. At the same time, the patients will need to imagine that the movements were performed by their affected arm and hand. In this group, only the non-affected arm and hand will need to perform the movements, but the affected one will not need to move.
  Arms: Uni-MVF condition and unimanual training mode using the new MT system (UM-UT)
Behavioral: Uni-MVF condition and bimanual training mode using the new MT system (UM-BT) — During the UM-BT, as similar as the first group (UM-UT), the participants will be also seated in front of the new MT system, and be instructed to watch the real-time image reflection of the non-affected arm and hand's movements on the screen carefully and imagine that the movements were performed by the affected arm. However, in this UM-BT group, the bilateral training mode is emphasized, and thus both arms and hands will need to move. That is, during therapy, the patient's affected arm and hand will be required to move at his/her best motor ability with the non-affected arm and hand at the same time.
  Arms: Uni-MVF condition and bimanual training mode using the new MT system (UM-BT)
Behavioral: Bi-MVF condition and bimanual training mode using the new MT system (BM-BT) — For the BM-BT group, the participants will be seated in front of this new MT system, and be instructed to observe the real-time image reflection of the non-affected arm and hand's movements transformed and superimposed on both arms and hands (i.e., bi-MVF), and to imagine that the movements were performed by both arms and hands. In this group, bi-MVF and bilateral training mode are emphasized, and thus both arms and hands will also need to move. The patient's affected arm and hand will be required to move as could as possible simultaneously.
  Arms: Bi-MVF condition and bimanual training mode using the new MT system (BM-BT)
Behavioral: Traditional MT using a mirror box — During traditional MT, the participants will be seated in front of a mirror box placed at their mid-sagittal plane. The affected arm and hand of the participants will be placed inside the mirror box, and the non-affected arm and hand will be in front of the mirror. As similar to the UM-UT group, the participants will be instructed to watch the mirror reflection of the movements performed by the non-affected arm and hand carefully and to imagine that the movements were performed by the aﬀected arm and hand. In this group, the patient's affected arm and hand inside the mirror box will not need to move.
  Arms: Traditional MT using a mirror box

SUMMARY:
The specific study aims will be:

1. To examine the treatment effects of a new digital mirror therapy (MT) system versus a mirror box in patients with stroke by conducting a 4-group randomized controlled trial.
2. To examine the electrophysiological mechanisms of uni-mirror visual feedback (uni-MVF) condition with unimanual training mode, uni-MVF condition with bimanual training mode, and bi-MVF condition with bimanual training mode in the new MT system by EEG.

DETAILED DESCRIPTION:
Part I: Validation of Treatment Efficacy of the New Digital MT System with Different MVF Conditions and Training Modes

In this new MT system, 3 different types of MT in different MVF conditions and training modes can be provided: unilateral MVF with unimanual training mode (UM-UT), unilateral MVF with bimanual training mode (UM-BT), and bilateral MVF with bimanual training mode (BM-BT). In the part Ⅰ study, an estimated total of 80 patients with stroke will be recruited. In addition to the original rehabilitation interventions of patients, each participant will be randomly allocated to 1 of 4 intervention groups (i.e., UM-UT, UM-BT, BM-BT, or traditional MT using a mirror box) for 15-hour therapy sessions. Outcome measures will be administrated at pre-treatment, immediately after treatment, and at 1-month follow-up after treatment.

Part II: Investigation of the Electrophysiological Mechanisms Underlying Different MVF Conditions by EEG

Twenty stroke patients will be recruited for examining the brain electrophysiological mechanisms underlying different types of MVF and training conditions of this new system by using electroencephalography (EEG). Three experimental conditions, including UM-UT, UM-BT, and BM-BT conditions, will be conducted in the EEG study.

ELIGIBILITY:
Part Ⅰ: Validation of Treatment Efficacy of the New Digital MT System with Different MVF Conditions and Training Modes

Inclusion Criteria:

* diagnosed with a unilateral stroke;
* at least 6 months after stroke onset;
* age between 20 and 80 years old;
* having a baseline score of Fugl-Meyer Assessment (FMA) in a range of 20 to 60;
* able to follow the study instructions;
* capable of participating in therapy and assessment sessions

Exclusion Criteria:

* global or receptive aphasia;
* severe neglect measured by line bisection test;
* other major medical diseases or comorbidities that have influenced upper-limb usage or caused severe pain

Part II: Investigation of the Electrophysiological Mechanisms Underlying Different MVF Conditions by EEG

Inclusion Criteria:

* diagnosed with a unilateral stroke;
* at least 2 weeks after stroke onset and medical stable;
* aged 20 to 80 years;
* having a baseline score of FMA ≥ 40 and wrist flexion ≥ 20 degrees in order to perform EEG motor tasks;
* both wrist flexion and extension scores of Modified Ashworth Scale ≤ 1;
* able to follow the study instructions

Exclusion Criteria:

* global or receptive aphasia;
* severe neglect measured by line bisection test;
* other major medical diseases or comorbidities, such as neurological and psychiatric diseases, that have caused severe pain of upper-limb or interfered brain neural activities

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Change scores of Fugl-Meyer Assessment | baseline (T0), at the end of 4 weeks of intervention (T1) , and 1 month after intervention (T2)
  The upper-limb subsection of Fugl-Meyer Assessment is a measure with sound psychometric properties to evaluate motor impairments.
Change scores of Chedoke Arm and Hand Activity Inventory | baseline (T0), at the end of 4 weeks of intervention (T1) , and 1 month after intervention (T2)
  The Chedoke Arm and Hand Activity Inventory is a reliable and validated measure to assess the independence of stroke patients to perform activities of daily living with an affected upper limb.

SECONDARY OUTCOMES:
change scores of Box and Block Test | baseline (T0), at the end of 4 weeks of intervention (T1) , and 1 month after intervention (T2)
  The Box and Block Test is a tool with sound reliability and validity to evaluate hand dexterity of stroke patients.
change scores of Revised Nottingham Sensory Assessment | baseline (T0), at the end of 4 weeks of intervention (T1) , and 1 month after intervention (T2)
  The Revised Nottingham Sensory Assessment is a standardized measure with good reliability to assess sensory function in patients with stroke.
change scores of Movement Imagery Questionnaire-Revised, Second Edition | baseline (T0), at the end of 4 weeks of intervention (T1) , and 1 month after intervention (T2)
  The Movement Imagery Questionnaire-Revised, Second Edition is a 14-item questionnaire with sound reliability and validity to evaluate the ability of motion imagination in patients with stroke.
change scores of Barthel Index | baseline (T0), at the end of 4 weeks of intervention (T1) , and 1 month after intervention (T2)
  The Barthel Index is a validated tool designed to measure activities reflecting the daily living independence.
change scores of Motor Activity Log | baseline (T0), at the end of 4 weeks of intervention (T1) , and 1 month after intervention (T2)
  The Motor Activity Log is a semi-structured interview with good psychometric properties to assess the level of use of affected upper limb in 30 main activities of daily living.
change scores of the health state of EQ-5D-5L | baseline (T0), at the end of 4 weeks of intervention (T1) , and 1 month after intervention (T2)
  The questionnaire of EQ-5D-5L contains 5 dimensions, including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and uses a 5-point Likert scale scored from 1 (no problem) to 5 (unable to/extreme problems); whereas, the numerical description of 5 dimensions represents the health state.
change scores of the visual analogue scale (VAS) of EQ-5D-5L | baseline (T0), at the end of 4 weeks of intervention (T1) , and 1 month after intervention (T2)
  The VAS of EQ-5D-5L scores will be scored from 0 to 100, with a higher score indicating better overall current health.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Wei Hsieh, PhD, Principal Investigator — Department of Occupational Therapy, College of Medicine, Chang Gung University
Locations (2):
- Taiwan (2):
  - Lo-Sheng Sanatorium and Hospital, Taoyuan, Taoyuan
  - Taoyuan Chang Gung Memorial Hospital, Taoyuan

IPD SHARING:
Plan to Share IPD: No